CLINICAL TRIAL: NCT02368418
Title: China Rural Health Initiative Follow up Study
Acronym: CRHIFU
Status: Completed | Type: Observational
Sponsor: The George Institute for Global Health, China (Other)
Responsible Party: Sponsor
Other Study IDs: PKU00001052
Record Dates: First submitted 2014-09-02; First posted 2015-02-23 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-01

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Rural health; China; Cohort study
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- PCP and SRS: participants had received two interventions (PCP and SRS)
  Interventions: Procedure: PCP; Procedure: SRS
- PCP only: participants had received PCP intervention only
  Interventions: Procedure: PCP
- SRS only: participants had received SRS intervention only
  Interventions: Procedure: SRS
- control group: participants had received usual care (neither PCP nor SRS)

INTERVENTIONS:
Procedure: PCP — PCP is short for the standard disease management program of individuals at high risk of cardiovascular disease delivered by Primary Care Providers (village doctors).
  Groups: PCP and SRS; PCP only
Procedure: SRS — SRS is short for a community-based Salt Reduction program delivered by community health educators.
  Groups: PCP and SRS; SRS only

SUMMARY:
China Rural Health Initiative (CRHI), a large-scale, factorial, cluster-randomized, controlled trial was conducted in 120 villages selected from 5 Northern Provinces of rural China between 2010 and 2012. Two interventions were evaluated through CRHI. One is the standard disease management program of individuals at high risk of cardiovascular disease delivered by Primary Care Providers (village doctors). Another one is a community-based Salt Reduction program delivered by community health educators. CRHI study interventions had ended for two years now and provide a good opportunity for us to understand whether its effects could be prolonged to a longer term. This study wants to evaluate the effects of CRHI interventions at 2 years after the end of CRHI (from Sep 2014 to Feb 2015).

In this follow-up survey, the baseline cohort of 5050 and post-intervention cohort of 4887 CRHI participants who were randomly selected from the 120 villages from 5 northern provinces of rural China will be recruited for the follow up study from Sep 2014 to Feb 2015. A questionnaire derived from CRHI baseline and post-intervention surveys will be used to collect data on disease history, medication use, care seeking patterns, lifestyle factors and so on. Weight, height, blood pressure and heart rate will be measured in the standard ways.

DETAILED DESCRIPTION:
"1."Background and Significance Cardiovascular disease (CVD) remains the number one global cause of death, accounting for 17.3 million deaths per year, a number that is expected to grow to 23.6 million by 2030. 80% of these deaths occur in low- and middle-income countries. These deaths were usually at younger ages compared to higher income countries.

CVD is the leading cause of death in China, responsible for approximately 3.5 million (41%) deaths in 2012. Reflecting the major contribution of cerebrovascular disease to the vascular disease burden in China, high blood pressure is the leading modifiable risk factor for cardiovascular disease and its importance is greatest in rural and northern regions where high blood pressure,salt consumption and the incidence of stroke are all very high.

Given the background above, China Rural Health Initiative, a large-scale, factorial, cluster-randomized, controlled trial was conducted in 120 villages selected from 5 Northern Provinces (Liaoning, Hebei, Shanxi, Shaanxi and Ningxia) of rural China between 2010 and 2012. CRHI aimed to develop, implement and evaluate effective, low-cost, and sustainable interventions for cardiovascular disease prevention and management suitable for widespread implementation in rural China. Two interventions were evaluated through CRHI. One is the standard disease management program of individuals at high risk of cardiovascular disease delivered by Primary Care Providers (village doctors) ('PCP' hereafter). Another one is a community-based Salt Reduction program delivered by community health educators ('SRS' hereafter).

A stratified randomization was used to assign the villages into 4 groups: PCP only, SRS only, both PCP and SRS, and usual care (neither PCP nor SRS). For the entire study, there were 60 villages with 'PCP' and 60 villages with 'no PCP' (with or without SRS) and 60 villages with 'SRS' and 60 villages with 'no SRS' (with or without PCP). For the PCP intervention, the period of intervention was 2 years; and for the SRS, approximately 1.5 years. And both interventions ended in November, 2012.

High risk individuals were defined as those meeting any one of the following criteria, regardless of current medication use:

* Physician-diagnosed history of coronary heart disease or stroke;
* Older age (50 years or older for men; 60 years or older for women - "50+/60+" hereafter) and having history of diabetes;
* Older age (50+/60+) and measured SBP≥160 mmHg A baseline and a post-intervention random sample surveys (2 independent samples) of older adults (50+/60+), 4800 each, were conducted in all of the 120 villages before and after the interventions for up to 10 and 12 weeks respectively. In each village at each survey, the survey collected data from 40 consenting age-eligible adults, half men and half women. As a matter of fact, 5050 and 4887 older adults had participated in the baseline and post-intervention surveys respectively.

The main results of CRHI showed that the SRS intervention significantly reduced sodium intake in intervention compared with control villages, and PCP intervention program significantly improved clinical care of the high risk patients in terms of the use of primary care, provision of lifestyle advice, use of antihypertensive treatment and use of aspirin.

Previous studies showed that life style and behavior interventions could have longer term effect after the end of the study that was designed to evaluate the interventions. For example, the Daqing study in China showed that intervention effects existed up to 14 years after the active intervention. The follow up of Trial of Hypertension Prevention (TOHP) I and II study participants, 10-15 years after the sodium reduction intervention trials, found that the risk of a cardiovascular event was 25% lower among those in the intervention group (relative risk 0.75, P=0.04), adjusted for trial, clinic, age, race, and sex. CRHI study interventions, SRS and PCP, had ended for two years now and provide a good opportunity for us to understand whether its effects could be prolonged to a longer term.

"2."Aims To evaluate the effects of CRHI interventions, both SRS and PCP, in 2 years after the end of CRHI.

"3."Study Design This is a cohort follow-up survey. The baseline cohort of 5050 and post-intervention cohort of 4887 CRHI participants who were randomly selected from the 120 villages from 5 northern provinces (Liaoning, Hebei, Shanxi, Shaanxi and Ningxia) of rural China will be recruited for the follow up study.

Except for those who died after the CRHI baseline or post-intervention surveys, all CRHI survey participants should be contacted and informed consent should be obtained. The reasons for not in contact or not in response should be documented.

A questionnaire derived from CRHI baseline and post-intervention surveys will be used to collect data on disease history, medication use, care seeking patterns, lifestyle factors and so on. Weight, height, blood pressure and heart rate will be measured in the standard ways.

The "train the trainers" model is used to train the survey interviewers. Only the interviewers who have passed the tests can participate in the field investigation.

The field investigation will be carried out from September 2014 to February 2015 in 5 Northern Provinces above. After confirming the identity and obtaining the informed consents from participants, interviewers will begin to collect information. The standard operating procedures will be developed and followed during the whole process.

Outcomes The primary outcomes will be mean systolic blood pressure level among all participants and those at high risk.

Secondary outcomes (among all participants and high-risk patients) include:

* Proportion of individuals regularly visiting the village clinic
* Proportion of individuals receiving lifestyle advice
* Proportion of individuals treated with a blood pressure lowering agent
* Proportion of individuals treated with aspirin
* Proportion of individuals having knowledge on salt reduction
* Proportion of individuals using low sodium salt
* Proportion of individuals adopting healthy behavior
* Proportion of individuals developing CVD event

"4."Quality control Intensive discussions on protocol and standard operating procedures were made during the design phase of the study. And only the interviewers who have passed the tests can participant in the field investigation. Moreover, all instruments including sphygmomanometers and weight scales will be purchased and calibrated centrally. In the investigation field, all interviewers will apply the standard questionnaire and follow the standard operating procedure. Double entry will be used for data entry and all analysis will be validated by an independent data analyst.

"5."Ethics review and human subject protection The project will be reviewed by the Ethics Committee of the Peking University Health Science Center in Beijing, China. Written consent will be obtained from all participants in the research. All participants will be free to quit from the study at any time with no explanation required. The risk of participating in the study is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Individuals had participated the baseline or post-intervention survey.

Exclusion Criteria:

* Death

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The baseline cohort of 5050 and post-intervention cohort of 4887 CRHI participants who were randomly selected from the 120 villages from 5 northern provinces (Liaoning, Hebei, Shanxi, Shaanxi and Ningxia) of rural China will be recruited for the follow up study.
Sampling Method: Probability Sample
Enrollment: 9164 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
mean systolic blood pressure level among all participants and those at high risk | from baseline and post-intervention to the follow up

SECONDARY OUTCOMES:
Proportion of individuals regularly visiting the village clinic among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals receiving lifestyle advice among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals treated with a blood pressure lowering agent among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals treated with aspirin among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals having knowledge on salt reduction among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals using low sodium salt among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals adopting healthy behavior among all participants and high-risk patients | from baseline and post-intervention to the follow up
Proportion of individuals developing CVD event among all participants and high-risk patients | from baseline and post-intervention to the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, PhD, Principal Investigator — The George Institute for Global Health, China
Locations (5):
- China (5):
  - Hebei Province Center for Disease Prevention and Control ,China, Shijiazhuang, Hebei
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - Ningxia Medical University School of Public Health, Yinchuan, Ningxia
  - Xi'an Jiaotong University, Xi'an, Shaanxi
  - Changzhi Medical College, China, Changzhi, Shanxi